CLINICAL TRIAL: NCT03962179
Title: VAC Stent: A Prospective Feasibility Study for the Treatment of Gastrointestinal Leakage Through a Combination of Covered Nitinol Stent and Negative Pressure Wound Treatment
Brief Title: Feasibility and Efficacy of a Combination of a SEMS and Vacuum Wound Treatment (VACStent)
Acronym: VACStent
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital of Cologne (Other)
Responsible Party: Principal Investigator, Seung-Hun Chon, PI, University Hospital of Cologne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-1053_1
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Perforation Esophagus; Esophageal Cancer; Esophageal Achalasia; Esophageal Diseases
Keywords: Perforation Esophagus, Esophageal Anastomotic Leak,
MeSH Terms: conditions — Esophageal Perforation; Esophageal Neoplasms; Esophageal Achalasia; Esophageal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VACStent Group (Experimental): Patient s who received a VACStent
  Interventions: Device: VACStent

INTERVENTIONS:
Device: VACStent — Evaluation of the suitability of the medical device for sealing leaks in the gastrointestinal tract

SUMMARY:
Open, prospective, one-arm feasibility and efficacy study of a European conformity (CE) certified Combination product of two CE certified medical devices in the intended indication.

Evaluation of the suitability of the medical device for sealing leaks in the gastrointestinal tract

DETAILED DESCRIPTION:
The investigators analyzed the outcome of using a hybrid medical device (self-expanding metal stents (SEMS) with negative pressure wound therapy) in the treatment of leaks of the upper gastrointestinal tract

ELIGIBILITY:
Inclusion Criteria:

* Patients with spontaneous, iatrogenic or postoperative leakage in the esophagus, evidence of leakage through an endoscopic examination
* Accessibility of the leak with the delivery system of the VAC stent

Exclusion Criteria:

* Simultaneous participation in other interventional exams
* Endoscopic inaccessibility of the affected section
* Full anticoagulation with international normalized ratio (INR) > 1.5 and / or partial thromboplastin time (PTT) > 50 sec, or platelets <20.000 / μl (after therapeutic correction an inclusion is possible)
* Unstable patients with severe septic disease, who have a clinical history
* Assessment an immediate operation for safe focus switch-off requires
* Ileus image with constant vomiting (after nasogastric tube and gastric emptying an inclusion possible)
* Persons who are in a dependency / employment relationship with the sponsor or examiner stand
* Accommodation in an institution for judicial or regulatory purposes arrangement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-22 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Technique - % of patients with successful implantation of VACStent | From date of first implantation of VACStent until the leak is sealed or the treatment is canceled from any serious medical cause, whichever came first, up to 12 months
  % of patients with successful implantation of VACStent

SECONDARY OUTCOMES:
Healing of leak - % of patients with successful implantation of VACStent | From date of first implantation of VACStent until the leak is sealed or the treatment is canceled from any serious medical cause, whichever came first, up to 12 months
  % of patients with a sealed leak after successful treatment with VACStent
Treatment of sepsis | From date of first implantation of VACStent until the leak is sealed or the treatment is canceled from any serious medical cause, whichever came first, up to 12 months
  % of patients with successful treatment of sepsis leak after successful implantation of VACStent
Migration rate | From date of first implantation of VACStent until the leak is sealed or the treatment is canceled from any serious medical cause, whichever came first, up to 12 months
  % of patients with migration of VACStent after successful implantation of VACStent
Bleeding | From date of first implantation of VACStent until the leak is sealed or the treatment is canceled from any serious medical cause, whichever came first, up to 12 months
  % of patients with bleeding after successful implantation of VACStent
Arrosion of tissue structures | From date of first implantation of VACStent until the leak is sealed or the treatment is canceled from any serious medical cause, whichever came first, up to 12 months
  % of patients with % of patients with bleeding after successful implantation of VACStent after successful treatment with VACStent
Sealing of leak - % of patients with successful implantation of VACStent | From date of first implantation of VACStent until the leak is sealed or the treatment is canceled from any serious medical cause, whichever came first, up to 12 months
  % of patients with a sealed leak after successful treatment with VACStent

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Hun Chon, M.D., Principal Investigator — University Hospital of Cologne
Locations (1):
- University Hospital of Cologne, Cologne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chon SH, Bartella I, Burger M, Rieck I, Goeser T, Schroder W, Bruns CJ. VACStent: a new option for endoscopic vacuum therapy in patients with esophageal anastomotic leaks after upper gastrointestinal surgery. Endoscopy. 2020 May;52(5):E166-E167. doi: 10.1055/a-1047-0244. Epub 2019 Dec 2. No abstract available. PMID 31791095
- [Derived] Chon SH, Scherdel J, Rieck I, Lorenz F, Dratsch T, Kleinert R, Gebauer F, Fuchs HF, Goeser T, Bruns CJ. A new hybrid stent using endoscopic vacuum therapy in treating esophageal leaks: a prospective single-center experience of its safety and feasibility with mid-term follow-up. Dis Esophagus. 2022 Apr 19;35(4):doab067. doi: 10.1093/dote/doab067. PMID 34561712